CLINICAL TRIAL: NCT02094625
Title: A Dose-Finding Study of N-Acetylcysteine (NAC) to Prevent Cisplatin-induced Hearing Loss in Children With Cancer
Brief Title: NAC to Prevent Cisplatin-induced Hearing Loss
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Etan Orgel, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-14-00270
Record Dates: First submitted 2014-03-13; First posted 2014-03-24 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Neuroectodermal Tumors, Primitive; Liver Neoplasms; Osteosarcoma; Other Childhood Cancers Using Cisplatin-based Regimens
Keywords: Cisplatin; N-acetylcysteine; Hearing Loss; Otoprotection
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive; Liver Neoplasms; Osteosarcoma; Hearing Loss | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetylcysteine Intervention (Experimental): This is a dose-finding study using a traditional 3+3 dose escalation scheme. Up to 18 subjects (3 dose levels as per below) will be enrolled to determine the maximum tolerated dose (MTD). The MTD is defined as per traditional 3+3 criteria of less than or equal to one dose-limiting toxicity at the dose level. Once the MTD is determined, subjects will be equally distributed at the "safe" dose levels (less than or equal to the MTD) to determine the optimum dose to achieve NAC levels in the blood necessary for hearing protection.
  As of August 2018: The dose-escalation phase was completed and dose-level three was selected for expansion in 9 subjects.
  Interventions: Drug: N-Acetylcysteine
- Observation only (No Intervention): Subjects who are ineligible to receive the study drug NAC will have the option to enroll for study assessments only including laboratory testing and hearing assessments identical to the experimental intervention arm. This is a "cohort of convenience" for which we anticipate up to 36 children will be enrolled over the course of the study.

INTERVENTIONS:
Drug: N-Acetylcysteine — NAC will be administered intravenously over ~60 minutes starting 4 hours following completion of cisplatin chemotherapy.
  Three dose levels have been pre-determined:
  Dose Level 1: 225 mg/kg Dose Level 2: 300 mg/kg Dose Level 3: 450 mg/kg
  Should Dose Level 3 exceed the MTD, the study will examine blood levels of NAC and if below the target blood level necessary for hearing protection, the study will "de-escalate" from Dose Level 3 to an intermediate Dose Level 2.5 and test a dose of 375 mg/kg.
  As of August 2018: Dose escalation completed with MTD not reached. Dose level 3 (450mg/kg) selected for expansion with NAC.
  Other Names: N-acteylcysteine; acteylcysteine injectable; Acetadote
  Arms: N-Acetylcysteine Intervention

SUMMARY:
Cisplatin is a key chemotherapy agent for the treatment of multiple childhood cancers but causes permanent hearing loss. This study investigates the drug N-acetylcysteine (NAC) to determine the dose necessary to protect hearing and also how well tolerated NAC is when combined with chemotherapy.

DETAILED DESCRIPTION:
The study is a dose-finding study of N-acetylcysteine (NAC) to protect hearing in children receiving cisplatin for the treatment of their cancer. NAC also has potential to protect the kidneys from cisplatin toxicity.

The study uses a 3+3 dose-escalation scheme to determine the dose of NAC necessary to achieve serum levels consistent with hearing protection in pre-clinical animal models. Three dose levels are predefined. Once the maximum tolerated dose is determined, an expansion cohort will then be enrolled to further evaluate tolerability as well as intra-patient and inter-patient variability in achieved serum levels. An option to enroll in a separate arm for study assessments only is available for those who do not wish to receive NAC. Hearing loss in the cohort will be assessed in the entire cohort in comparison to historical and non-treated children to evaluate for trends toward efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Are between 1 and 21 years of age (inclusive) at time of diagnosis of underlying malignancy
* Have a new diagnosis of a localized malignancy with a planned treatment course to include at least two cycles of cisplatin
* Diagnosis to be assigned by oncology attending of record (may be reported via designee), histological diagnosis does not need to be confirmed separately
* Most common but not exclusive diagnoses consist of hepatoblastoma, medulloblastoma, osteosarcoma
* Total cumulative dose of planned cisplatin must be >200 mg/m2 (or 6.67 mg/kg equivalent for infants requiring weight-based dosing. Conversion factor used is 30:1).
* Cisplatin must be delivered over <3 days
* Planned cisplatin dose to be infused over ≤6 hours for ≤2 days per cycle
* Are anticipated to be able to comply with end-of-therapy audiology assessment (note that hearing assessments are performed per routine clinical care in children receiving cisplatin and consist of an audiogram or auditory brainstem response, and distortion-product otoacoustic emissions)
* Patients with any hearing status are eligible for study (as long as they can comply with the study primary aims of assessing toxicity and dose-response)

Exclusion Criteria:

* no preexisting risk of serious arrhythmia as defined by (a) normal sinus rhythm on electrocardiogram and corrected QT interval <500 and (b) no previous history of congenital arrhythmia (e.g. Wolf-Parkinson-White)
* Hepatic, biliary, cardiac, or bone marrow function inadequate for chemotherapy as per patient's treatment regimen. There are no additional protocol-specific restrictions for these markers.
* Moderate or Severe Persistent Asthma as defined by the latest recommendations from the National Heart Lung and Blood Institute definition includes daily asthma exacerbation with need for rescue medication) or an overnight hospitalization for asthma exacerbation within the previous 28 days
* Disseminated disease (e.g. lepto-meningeal spread, tumor metastases)
* Karnofsky or Lansky score <50%
* Pregnancy or breast-feeding mothers
* Documented hypersensitivity or allergy to previous NAC infusion

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Target Serum Level NAC | On average up to 4 weeks from diagnosis
  Following the first dose of cisplatin, NAC will be administered as described below. A NAC level will then be measured immediately following this first dose of NAC to determine if the blood (serum) level reaches the threshold necessary for hearing protection.

SECONDARY OUTCOMES:
Adverse events during infusion of NAC | Up to approximately 40 weeks from start of chemotherapy (regimen dependent)
  Subjects will be monitored during and after each NAC infusion to determine how well they tolerate the drug. Infusion rate related and spontaneously resolving "anaphylactoid" reactions are the most common reported toxicity and will be closely monitored. Most subjects will receive 3 cycles of cisplatin and NAC, typically within the first 15 weeks of starting chemotherapy. Subjects who continue to receive cisplatin and NAC for additional cycles will continue to be monitored.
NAC Level | -6,0, 0.5, and 4 hours from start of first NAC dose (intervention)
  A NAC serum level will be measured surrounding the first dose of NAC at 4 times:
  1. pre-cisplatin (baseline)
  2. following cisplatin/before NAC
  3. immediately following NAC (primary aim)
  4. delayed four hours following NAC
  For those in the non-intervention arm, NAC serum levels will be measured at corresponding times as determined by the start of the cisplatin infusion.
Hearing assessment | Up to approximately 40 weeks from start of chemotherapy
  Routinely performed hearing assessments will be analyzed at the end of therapy as compared to a historical cohort, non-treated, and to patient's baseline (if available) to evaluate for any trend toward a protective effect from NAC.
Renal Toxicity | Up to approximately 40 weeks from start of chemotherapy
  Information regarding renal toxicity due to cisplatin will be collected at end of therapy and compared to historical rates and non-treated patients to evaluate a potential protective effect by NAC
Response of tumor to treatment | On average up to 15 weeks from start of chemotherapy (regimen dependent)
  Early indicators of tumor response to cisplatin-based chemotherapy (e.g. percent necrosis in resected tumors, early remission rates, etc) will be informally evaluated in comparison to historical data for any evidence NAC decreases efficacy of the chemotherapy
Effect of Genotype on Hearing Loss and Hearing Protection | On average up to 15 weeks from start of chemotherapy
  Saliva/cheek swabs will be collected one-time for genotype analysis to examine the influence of glutathione polymorphisms on cisplatin-induced hearing loss and NAC hearing protection
Glutathione serum level | -6,0, 0.5, and 4 hours from start of first NAC dose (intervention)
  Glutathione serum levels will be measured at times corresponding to NAC levels surrounding the first dose of NAC at 4 times:
  1. pre-cisplatin (baseline)
  2. following cisplatin/before NAC
  3. immediately following NAC (primary aim)
  4. delayed four hours following NAC
  For those in the non-intervention arm, serum levels will again be measured at corresponding times as determined by the start of the cisplatin infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Etan Orgel, MD MS, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States